CLINICAL TRIAL: NCT00295360
Title: Influence of Cholestasis on Intestinal BCRP Expression
Brief Title: Expression of BCRP in Icteric Patients
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Other Study IDs: MDR-108-03
Record Dates: First submitted 2006-02-17; First posted 2006-02-23 (Estimated); Last update posted 2006-02-23 (Estimated); Status verified 2005-03

CONDITIONS: Icterus
Keywords: cholestasis; BCRP; multidrug resistance; duodenum; bile acids; ABCG2
MeSH Terms: conditions — Jaundice; Cholestasis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Behavioral: no intervention, pathophysiological study

SUMMARY:
The expression of transporters involved in bile acid homeostasis is differentially regulated during obstructive cholestasis. Bile acids are also substrates of the drug efflux transporter breast cancer resistance protein (BCRP) that is highly expressed in the human intestine. Therefore we intend to analyze whether intestinal BCRP expression could be altered during cholestasis.

DETAILED DESCRIPTION:
BCRP is capable of transport bile acids and may indicate that this transporter is involved in bile acid homeostasis. As an efflux pump, it could protect the enterocytes from potential toxic bile acid concentrations. During cholestasis, where the enterohepatic circulation is disrupted, there occurs an adaptive regulation of transporters for bile acids, bilirubin and cholesterol. These changes take place in liver, kidney, as well as in the intestine.

Using real-time RT-PCR analysis we determine BCRP mRNA expression levels in duodenal tissue of healthy subjects and cholestatic patients. BCRP protein levels will be determined by immunohistochemistry.

Healthy subjects and cholestatic patients are enrolled in the study after giving informed consent. Control subjects with an indication for a gastrointestinal tract endoscopy within a cancer-screening program and patients with obstructive cholestasis with an interventional endoscopic retrograde cholangiopancreatography (ERCP) are included in this study. During endoscopy four biopsy specimens are obtained from the distal part of the duodenum. Biopsies are immediately stored at -70°C until further processing.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of obstructive cholestasis (obstructive jaundice was defined on the basis of chemical parameters (bilirubin, g-glutamyltransferase, and alkaline phosphatase) and on imaging procedures (ultrasound and ERCP) demonstrating a dilated bile duct system)
* control subjects had an indication for a gastrointestinal tract endoscopy within a cancer-screening program

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2003-06; Study Completion 2004-08

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Drewe, MD, MSc, Principal Investigator — Department of Clinical Pharmacology, University Basel
Locations (1):
- University Basel, Department of Research, Basel, Canton of Basel-City, Switzerland